CLINICAL TRIAL: NCT00803595
Title: A Randomized Double-blind Controlled Study of CS-8958 Versus Oseltamivir Phosphate in Patients With Influenza Virus Infection
Brief Title: A Multinational Phase III Study of CS-8958 (MARVEL)
Acronym: MARVEL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Daiichi Sankyo Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Daiichi Sankyo (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CS8958-A-J301
Record Dates: First submitted 2008-12-04; First posted 2008-12-05 (Estimated); Results first posted 2011-11-22 (Estimated); Last update posted 2019-01-09 (Actual); Status verified 2011-11

CONDITIONS: Influenza, Human
Keywords: Influenza; Neuraminidase inhibitor
MeSH Terms: conditions — Influenza, Human | interventions — CS 8958; Oseltamivir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- CS-8958 Low Dose (Experimental): CS-8958 powder to be inhaled - low-dose arm
  Interventions: Drug: CS-8958
- CS-8958 High Dose (Experimental): CS-8958 powder to be inhaled - high-dose arm
  Interventions: Drug: CS-8958
- Oseltamivir phosphate (Active Comparator): oseltamivir phosphate oral capsules
  Interventions: Drug: oseltamivir phosphate

INTERVENTIONS:
Drug: CS-8958 — CS-8958 powder 20 mg to be inhaled one time. Oseltamivir phosphate placebo capsules 2 times per day for 5 days
  Arms: CS-8958 Low Dose
Drug: CS-8958 — CS-8958 powder 40 mg to be inhaled one time. Oseltamivir phosphate placebo capsules 2 times per day for 5 days
  Arms: CS-8958 High Dose
Drug: oseltamivir phosphate — CS-8958 placebo powder to be inhaled one time. Oseltamivir phosphate oral capsules taken twice daily for 5 days.
  Arms: Oseltamivir phosphate

SUMMARY:
The primary objective of this study is to confirm the efficacy of CS-8958 administered as a single inhaled low dose or single inhaled high dose by showing non-inferiority to oseltamivir phosphate using the time to alleviation of influenza illness. For safety evaluation, between-group comparisons will be made with regard to incidence of adverse events and other safety measures.

In a secondary objective, the optimum dosage of CS-8958 for this indication will be evaluated based on the efficacy and safety of single inhaled low or high dose.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of influenza
* Axillary temperature of > or = to 37.5 degrees C

Exclusion Criteria:

* Infection by bacteria species and/or virus other than influenza virus
* Chronic respiratory disease
* Renal dysfunction

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1002 (Actual)
Dates: Start 2008-11; Primary Completion 2009-03 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- Hong Kong, China
- Tokyo, Japan
- Seoul, South Korea
- Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

REFERENCES:
- [Derived] Watanabe A, Chang SC, Kim MJ, Chu DW, Ohashi Y; MARVEL Study Group. Long-acting neuraminidase inhibitor laninamivir octanoate versus oseltamivir for treatment of influenza: A double-blind, randomized, noninferiority clinical trial. Clin Infect Dis. 2010 Nov 15;51(10):1167-75. doi: 10.1086/656802. Epub 2010 Oct 11. PMID 20936975

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This multicenter, double-blind,randomized, active-controlled trial was conducted from November 2008 through March 2009 at 117 institutions in Japan, Taiwan, Korea, and China (Hong Kong).
Pre-assignment Details: Full analysis set (FAS) was defined as the set of subjects who had a positive test result using the influenza rapid diagnostic kit, received at least 1 dose of the study drug, and had valid efficacy data. The data for the baseline characteristics is provided for this analysis set, not for all participants who entered the trial.
Groups:
- CS-8958 High Dose 40 mg: CS-8958 powder to be inhaled - high-dose arm
- CS-8958 Low Dose 20 mg: CS-8958 powder to be inhaled - low-dose arm
- Oseltamivir 75 mg: oseltamivir phosphate oral capsules
Period: Overall Study
Arm/Group | CS-8958 High Dose 40 mg | CS-8958 Low Dose 20 mg | Oseltamivir 75 mg
Started | 337 | 327 | 338
Completed | 322 | 319 | 322
Not Completed | 15 | 8 | 16
Not completed — Adverse Event | 3 | 4 | 1
Not completed — Protocol Violation | 7 | 2 | 12
Not completed — Withdrawal by Subject | 5 | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CS-8958 High Dose 40 mg | CS-8958 Low Dose 20 mg | Oseltamivir 75 mg | Total
Number analyzed (Participants) | 334 | 326 | 336 | 996
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.9 (11.5) | 35.6 (11.7) | 34.7 (11.3) | 35.0 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 155 | 164 | 158 | 477
  Male | 179 | 162 | 178 | 519
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 334 | 326 | 336 | 996
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Taiwan | 62 | 61 | 63 | 186
  China | 3 | 2 | 2 | 7
  Japan | 263 | 256 | 266 | 785
  Korea, Republic of | 6 | 7 | 5 | 18
Laboratory confirmed influenza [Number; unit: Participants]
  Virus A/H1N1 | 218 | 215 | 212 | 645
  Virus A/H3N2 | 108 | 102 | 112 | 322
  Virus B | 0 | 2 | 1 | 3
  Negative | 8 | 7 | 11 | 26

OUTCOME MEASURES:

1. Primary Outcome: Time to Alleviation of Influenza Illness
Description: The time to illness alleviation which was defined as the time from the initiation of trial treatment to the beginning of the first 21.5-h period in which all influenza symptoms were "absent" or "mild." Patients recorded their severity of influenza symptoms (headache, myalgia/arthralgia, fatigue, chills/sweats, nasal symptom, sore throat, and cough) 4 times daily for 15 days. Patients whose influenza symptoms had not been alleviated at the time of their withdrawal from the study or at the end of the observation period were censored.
Time Frame: 15 days
Population: Full analysis set (FAS) was defined as the set of subjects who had a positive test result using the influenza rapid diagnostic kit, received at least 1 dose of the study drug, and had valid efficacy data.
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | CS-8958 High Dose 40 mg | CS-8958 Low Dose 20 mg | Oseltamivir 75 mg
Number analyzed (Participants) | 334 | 326 | 336
hours | 73.0 [68.4 to 80.8] | 85.8 [76.5 to 92.8] | 73.6 [68.5 to 83.3]
Statistical Analysis 1: Comparison: CS-8958 Low Dose 20 mg vs Oseltamivir 75 mg; This trial was designed to confirm the efficacy of laninamivir octanoate by showing that the median time to illness alleviation in patients treated with laninamivir octanoate was not >18 hours longer than that in patients treated with oseltamivir. Sample size of 300 patients in each group was determined to achieve a power of at least 80% to show noninferiority at both dose levels of laninamivir octanoate with use of a Monte Carlo simulation; Test type: Non-Inferiority or Equivalence — A noninferiority margin of 18 hours (h) was set to assure the superiority of laninamivir octanoate over a putative placebo. A meta-analysis using 3 placebo-controlled trials reported that the difference between the median time to illness alleviation in the placebo and oseltamivir groups was 33.1 h and the 95% confidence interval ranged from 19.1 to 47.1 h. From this, a margin that was less than the lower limit of this 95% CI was selected; p = 0.748, Generalized Wilcoxon Test — 2-sided p-value without adjustments for multiple testing; Median Difference (Final Values) = -0.6, 95% CI 2-sided [-9.9 to 6.9]
Statistical Analysis 2: Comparison: CS-8958 High Dose 40 mg vs CS-8958 Low Dose 20 mg; Null hypothesis was that there was no difference in the time to illness alleviation; Test type: Superiority or Other; p = 0.038, Generalized Wilcoxon Test — 2-sided p-value without adjustments for multiple testing; Median Difference (Final Values) = -12.8, 95% CI 2-sided [-18.2 to -0.4]
Statistical Analysis 3: Comparison: CS-8958 Low Dose 20 mg vs Oseltamivir 75 mg; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — A noninferiority margin of 18 hours was set to assure the superiority of laninamivir octanoate over a putative placebo. A meta-analysis using 3 placebo-controlled trials reported that the difference between the median time to illness alleviation in the placebo and oseltamivir groups was 33.1 h and the 95% confidence interval ranged from 19.1 to 47.1 h. From this, a margin that was less than the lower limit of this 95% CI was selected; p = 0.104, Generalized Wilcoxon test; Median Difference (Final Values) = 12.2, 95% CI 2-sided [-1.5 to 17.2]

2. Secondary Outcome: Time for Body Temperature to Return to Normal
Description: Time for return to normal axillary temperature was was defined as the time until the beginning of the first 21.5-hour period in which the axillary temperature returned to 36.9°C. Patients recorded their axillary temperature 4 times daily for 15 days. Patients whose axillary temperature had not been returned to 36.9°C at the time of their withdrawal from the study or at the end of the observation period were censored.
Time Frame: 15 days
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | CS-8958 High Dose 40 mg | CS-8958 Low Dose 20 mg | Oseltamivir 75 mg
Number analyzed (Participants) | 334 | 326 | 336
hours | 55.3 [46.6 to 64.0] | 58.0 [52.3 to 66.9] | 54.7 [48.2 to 62.2]
Statistical Analysis 1: Comparison: CS-8958 Low Dose 20 mg vs Oseltamivir 75 mg; Null hypothesis was that there was no difference in the time for return to normal axillary temperature; Test type: Superiority or Other; p = 0.318, Generalized Wilcoxon test — 2-sided P value without adjustments for multiple testing; Median Difference (Final Values) = 3.3, 95% CI 2-sided [-2.8 to 9.1]
Statistical Analysis 2: Comparison: CS-8958 High Dose 40 mg vs Oseltamivir 75 mg; Null hypothesis was that there was no difference in the time for return to normal axillary temperature; Test type: Superiority or Other; p = 0.981, Generalized Wilcoxon test — 2-sided P value without adjustments for multiple testing; Median Difference (Final Values) = 0.6, 95% CI 2-sided [-5.8 to 5.7]
Statistical Analysis 3: Comparison: CS-8958 High Dose 40 mg vs CS-8958 Low Dose 20 mg; Null hypothesis was that there was no difference in the time for return to normal axillary temperature; Test type: Superiority or Other; p = 0.344, Generalized Wilcoxon test — 2-sided P value without adjustments for multiple testing; Median Difference (Final Values) = -2.7, 95% CI 2-sided [-9.1 to 3.1]

ADVERSE EVENTS:
Time Frame: 15 days
Arm/Group | CS-8958 High Dose 40 mg | CS-8958 Low Dose 20 mg | Oseltamivir 75 mg
Serious Adverse Events (participants affected / at risk) | 0/337 | 0/326 | 2/336
Other Adverse Events (participants affected / at risk) | 63/337 | 54/326 | 63/336
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CS-8958 High Dose 40 mg (N=337) | CS-8958 Low Dose 20 mg (N=326) | Oseltamivir 75 mg (N=336)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Wallenberg syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CS-8958 High Dose 40 mg (N=337) | CS-8958 Low Dose 20 mg (N=326) | Oseltamivir 75 mg (N=336)
Diarrhoea (Gastrointestinal disorders) | 26 | 18 | 26
Nausea (Gastrointestinal disorders) | 4 | 7 | 6
Vomiting (Gastrointestinal disorders) | 1 | 1 | 8
Gastroenteritis (Infections and infestations) | 4 | 0 | 0
Nasopharyngitis (Infections and infestations) | 12 | 3 | 8
Oral herpes (Infections and infestations) | 2 | 3 | 4
Alanine aminotransferase increase (Investigations) | 5 | 4 | 2
Platelet count increased (Investigations) | 3 | 6 | 1
Dizziness (Nervous system disorders) | 3 | 6 | 0
Headache (Nervous system disorders) | 1 | 3 | 4
Urticaria (Skin and subcutaneous tissue disorders) | 2 | 3 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principle investigator shall not publish the results of the study at any time without the prior written approval of Sponsor.